CLINICAL TRIAL: NCT03988816
Title: Effect of Roflumilast on Quality of Life, Lung Function and Mucus Properties in Patients With Non-cystic Fibrosis Bronchiectasis: a Cross-over, Unicentric, Double-blind and Placebo-controlled Study
Brief Title: Effect of Roflumilast on Quality of Life, Lung Function and Mucus Properties in Patients With Bronchiectasis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SDC 4706/18/057; 2018/17035-5 (Other Grant/Funding Number: FAPESP)
Record Dates: First submitted 2019-06-14; First posted 2019-06-17 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-06

CONDITIONS: Bronchiectasis Adult
Keywords: bronchiectasis; lung function; quality of life; mucus properties
MeSH Terms: conditions — Bronchiectasis | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Roflumilast (Experimental): Roflumilast tablets will be supplied at a concentration of 500 mcg. Each tablet contains 500mcg of the active ingredient in addition to the excipients: lactose monohydrate, corn starch, povidone and magnesium stearate. The coating contains hypromellose, macrogol, titanium dioxide, yellow iron oxide. Patients should take 1 tablet once daily, before, during or after meals, at the same time each day.
  Interventions: Drug: Roflumilast
- Placebo (control) (Placebo Comparator): Roflumilast placebo-containing tablets will look similar to active roflumilast tablets and will be supplied to patients in packs identical to those of the active drug.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Roflumilast — 500Mcg Tab, once daily
  Other Names: Daxas
  Arms: Roflumilast
Drug: Placebo oral tablet — once daily
  Other Names: Placebo
  Arms: Placebo (control)

SUMMARY:
Although relatively common, bronchiectasis is considered an orphan disease as there is little evidence for adequate treatment, most of the therapeutic options are extrapolated from studies with patients with chronic obstructive pulmonary disease (COPD) or cystic fibrosis (CF). Inhaled bronchodilators and corticosteroids should be used as a therapeutic test and maintained if there is improvement of symptoms or lung function. There is no evidence to justify the use of mucolytic agents for these patients. The treatment with greater evidence is the use of macrolides, especially azithromycin. A meta-analysis published in 2014 showed that there was a reduction in the number of exacerbations, an improvement in the quality of life and a reduction in the decrease in FEV1. However, studies have shown conflicting results regarding quality of life and pulmonary function.

Roflumilast is a phosphodiesterase-4 inhibitor with an anti-inflammatory effect in vitro and in vivo due to the inhibition of cyclic adenosine monopostat breakdown (cAMP) to its inactive phosphodiesterase form. As this enzyme is expressed in high concentrations in leukocytes and other inflammatory cells responsible for the pathogenesis of pulmonary diseases such as COPD, it has been studied and used for this disease. COPD is characterized by a chronic inflammatory process of the airways, predominantly neutrophils and high levels of proinflammatory cytokines related to this cell, such as interleukin-8, neutrophil elastase, tumor necrosis factor (TNF) alpha and E-selectin. The REACT study showed that roflumilast prevents moderate and severe infectious exacerbations in addition to improved lung function in patients with COPD who continue to exacerbate despite the use of combined bronchodilator and inhaled corticosteroid therapy.

Since bronchiectasis and COPD are chronic inflammatory diseases, they present similar inflammatory processes, with neutrophil as the main inflammatory cell, it is expected that the use of roflumilast also has an anti-inflammatory effect in bronchiectasis. In addition, since bronchiectasis is a disease with poor evidence for pharmacological treatment, it is necessary to search for new therapeutic possibilities.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* Diagnosis of bronchiectasis by chest tomography;
* FEV1 <60% of predicted;
* History of chronic bronchitis (chronic cough and sputum for at least 3 months in the last 2 years);
* 2 or more infectious exacerbations in the last year (defined as worsening of cough and / or dyspnoea and / or decreased general condition, increased quantity and purulence of sputum that required systemic antibiotic use (oral or intravenous).

Exclusion Criteria:

* Hemoptysis in the last 6 months (significance at the discretion of the investigator);
* Current or prior smoking if > 10 pack-years;
* FEV1 < 30% of predicted;
* Known allergy to roflumilast;
* Pulmonary exacerbation present or occurring in the last 4 weeks;
* Child B or C cirrhosis;
* Active cancer (except basal cell carcinoma);
* Severe heart failure;
* Depression associated with suicidal ideation;
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-12-06 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life questionnaire | 12 weeks
  To evaluate the impact of roflumilast on the quality of life of patients with bronchiectasis through the Saint George Respiratory Questionnaire (SGRQ).

SECONDARY OUTCOMES:
Other tools for quality of life | 12 weeks
  To evaluate the impact of roflumilast on quality of life using the questionnaires Leicester, Quality of Life Questionnaire-Bronchiectasis (QOL-B) Bronchiectasis Health Questionnaire (BHQ)
Dyspnea | 12 weeks
  To evaluate the impact of roflumilast on severity of dyspnea as measured by the COPD Assessment Test (CAT)
Lung function | 12 weeks
  To evaluate the impact of roflumilast on lung function measured by forced expiratory volume at one second (FEV1)
Adverse events | 12 weeks
  To evaluate the safety of roflumilast assessed through the incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo A Athanazio, MD, PhD, Principal Investigator — Medical Assistant
Locations (1):
- Heart Institute (InCor) - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fjaellegaard K, Sin MD, Browatzki A, Ulrik CS. Antibiotic therapy for stable non-CF bronchiectasis in adults - A systematic review. Chron Respir Dis. 2017 May;14(2):174-186. doi: 10.1177/1479972316661923. Epub 2016 Aug 9. PMID 27507832
- [Background] Quint JK, Millett ER, Joshi M, Navaratnam V, Thomas SL, Hurst JR, Smeeth L, Brown JS. Changes in the incidence, prevalence and mortality of bronchiectasis in the UK from 2004 to 2013: a population-based cohort study. Eur Respir J. 2016 Jan;47(1):186-93. doi: 10.1183/13993003.01033-2015. Epub 2015 Nov 5. PMID 26541539
- [Background] McShane PJ, Naureckas ET, Tino G, Strek ME. Non-cystic fibrosis bronchiectasis. Am J Respir Crit Care Med. 2013 Sep 15;188(6):647-56. doi: 10.1164/rccm.201303-0411CI. PMID 23898922
- [Background] Beghe B, Rabe KF, Fabbri LM. Phosphodiesterase-4 inhibitor therapy for lung diseases. Am J Respir Crit Care Med. 2013 Aug 1;188(3):271-8. doi: 10.1164/rccm.201301-0021PP. PMID 23656508
- [Background] Grootendorst DC, Gauw SA, Verhoosel RM, Sterk PJ, Hospers JJ, Bredenbroker D, Bethke TD, Hiemstra PS, Rabe KF. Reduction in sputum neutrophil and eosinophil numbers by the PDE4 inhibitor roflumilast in patients with COPD. Thorax. 2007 Dec;62(12):1081-7. doi: 10.1136/thx.2006.075937. Epub 2007 Jun 15. PMID 17573446